CLINICAL TRIAL: NCT01041495
Title: An Eight Week, Double-Blind Efficacy Study of Cyclobenzaprine ER (Amrix TM) Augmentation to Alleviate Fibromyalgia Fatigue and Muscle Pain
Brief Title: Cyclobenzaprine Extended Release (ER) for Fibromyalgia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: ran out of funding short of enrollment expected
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Cephalon, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas L. Schwartz, M.D., Assoc Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: amrixfm001
Record Dates: First submitted 2009-06-29; First posted 2009-12-31 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia; Pain; Sleep; Fatigue
Keywords: fibromyalgia; Pain; Sleep; Fatigue
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue | interventions — cyclobenzaprine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cyclobenzaprine ER (Experimental): active drug
  Interventions: Drug: cyclobenzaprine ER (AMRIX)
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cyclobenzaprine ER (AMRIX) — active drug
  Other Names: AMRIX
  Arms: cyclobenzaprine ER
Drug: placebo — matching placebo for cyclobenzaprine ER (AMRIX)
  Other Names: matching placebo for cyclobenzaprine ER (AMRIX)
  Arms: placebo

SUMMARY:
Amrix (Cyclobenzaprine hydrochloride Extended release capsules) is approved by the FDA as a muscle relaxant, indicated for the treatment of muscle spasm associated with acute, painful musculoskeletal conditions. Cyclobenzaprine ER (Amrix TM) has a distinct pharmacokinetic profile providing early systemic exposure and consistent plasma concentration over several hours. Overall, a single dose of Amrix 30 mg is similar to that of cyclobenzaprine immediate release 10 mg three times daily. This ER formula should improve compliance, with similar efficacy and possibly less side effects as is often the case with slower release formulations.

There are clinical studies showing that cyclobenzaprine can alleviate pain secondary to Fibromyalgia induced muscle tone. This multi-layered evidence base suggests that cyclobenzaprine may be able to alleviate pain in fibromyalgia. Theoretically in fibromyalgia, pain is interpreted centrally and possibly occurs due to said muscle spasm . Cyclobenzaprine may relieve this pain, thus allowing patients to function better during the day and sleep better at night. Cyclobenzaprine has tricyclic antidepressant structure which may also allow pain signal dampening in the spinal cord as well, similar to amitriptyline which is used off-label for neuropathic pain as well.

Fibromyalgia (FM) is an illness that may involve medical, rheumatologic, autoimmune, sleep, endocrine and psychiatric pathology. It is a syndrome of recurrent pain at trigger points. Greater than 90% of these patients will report fatigue as a key symptom as well. There are several investigation lines into the treatment of FM induced pain. Exercise, behavioral therapy, amitryptiline, duloxetine, tramadol, sodium oxybate, pregabalin all have randomized trials and almost all focus on pain. There are very few studies evaluating cyclobenzaprine and none studying to Cyclobenzaprine ER formulation. None evaluate pain reduction, sleep and fatigue improvement.

Cyclobenzaprine is a drug with minimal adverse effects (dry mouth, dizziness, fatigue, constipation, somnolence, nausea, and dyspepsia). It may have a safer tolerability profile than some of the FM medications noted above. As cyclobenzaprine is often studied and often added as an augmentation agent to patients' regimens who suffer from acute painful musculoskeletal conditions, the authors feel that cyclobenzaprine would also be effective in this population. The authors wish to conduct a study to determine if cyclobenzaprine ER is safe and tolerable in the treatment of FM induced pain, and secondary fatigue and insomnia. This initial study may allow for continued regulatory studies with this product in FM subjects. The authors propose a double-blind placebo controlled study to determine if cyclobenzaprine ER is safe and effective in reversing FM induced pain, and secondary fatigue and insomnia.

ELIGIBILITY:
Inclusion Criteria:

If possible, 60 subjects will be included in this study.

* All males/females of any race are eligible if aged between 18 and 65 and
* Subjects must speak English and have capacity to receive and utilize informed consent
* Agree to use barrier method contraception or are infertile x 2 years due to medical condition or surgery
* Have been formally diagnosed by a Board Certified Rheumatologist using the ACR 1990 research criteria for fibromyalgia
* Report that pain is a key distressing symptom of their FM
* Have a score of > 4 on the Visual Analogue Pain Scale (VAPS)

Exclusion Criteria: Subjects cannot

* Be pregnant or be attempting to conceive at present (urine bHCG must be negative)
* Have an active substance abuse problem with last use within the past 90 days (outside of nicotine)
* Use cardiac QTc prolonging medications i.e., tricyclic antidepressants
* Use p4502D6 major inhibiting medications as cyclobenzaprine levels may increase
* Have a known medical condition outside of FM that causes pain, i.e., diabetic neuropathy
* Have a known medical condition or other medication use that relatively contraindicates cyclobenzaprine use (i.e., hypersensitivity concomitant use of monoamine oxidase (MAO) inhibitors, seizures, known cardiac abnormalities, recent MI. hepatitis, stroke, or psychosis
* Has a prior history of cyclobenzaprine use and failure (failure due to side effects may be allowed at P.I. discretion)
* Be receiving daytime/nighttime sedating medication with clear chronological impact on fatigue UNLESS fatigue predates sedating medication or said medication has been steadily dosed > 4 weeks
* Other medications known to alleviate pain (i.e., Gabapentin, Pregabalin, Amitryptiline, Duloxetine,Venlafaxine, Carbamazepine, Tramadol, etc) unless they have been at steady dose more than 6 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: thomas l schwartz, md, Principal Investigator — SUNY Upstate
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: radio and billboard ads were used to recruit subjects who were then screened a a psychiatric based practice
Pre-assignment Details: subjects had to meet eligibility criteria
Groups:
- Cyclobenzaprine ER: active muscle relaxant medication
- Placebo: matching placebo
Period: Overall Study
Arm/Group | Cyclobenzaprine ER | Placebo
Started | 16 | 12
Completed | 12 | 5
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclobenzaprine ER | Placebo | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Pain Scale at 8 Weeks Post Treatment
Description: Visual Analogue Pain Scale -Change in baseline subjective pain based on a 10 point scale (1= no pain, 10 = severe pain) from baseline (T=Zero, prior to drug/placebo treatment) to week 8. Higher scores are worse
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Placebo: placebo: matching placebo for AMRIX
Arm/Group | Cyclobenzaprine ER | Placebo
Number analyzed (Participants) | 16 | 12
units on a scale | 4.8 [4 to 6] | 5.7 [5 to 6]
Statistical Analysis 1: Comparison: Cyclobenzaprine ER vs Placebo; Test type: Superiority or Other; p = .869, t-test, 2 sided — P values below 0.05 were considered statistically significant; Mean Difference (Final Values) = .869

2. Secondary Outcome: Brief Fatigue Inventory at 8 Weeks Post Treatment
Description: Brief Fatigue Inventory- Change in baseline subjective fatigue based on this scale (1= no fatigue, 10 = severe fatigue) from baseline (T=Zero, prior to drug/placebo treatment) to week 8 where higher scores are worse
Time Frame: baseline to 8 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cyclobenzaprine ER | Placebo
Number analyzed (Participants) | 16 | 12
score on a scale | 4.7 [4 to 6] | 4.8 [4 to 5]
Statistical Analysis 1: Comparison: Cyclobenzaprine ER vs Placebo; Visual Analogue Pain Scale (VAPS). The final visit VAPS at 8th week will be compared against baseline VAPS scores for both treatment groups; Test type: Superiority or Other; p = .486, t-test, 2 sided; Mean Difference (Final Values) = 4
Statistical Analysis 2: Comparison: Cyclobenzaprine ER vs Placebo; Test type: Superiority; p = .486, t-test, 1 sided; Mean Difference (Final Values) = 1

3. Secondary Outcome: Fibromyalgia Impact Questionnaire Scores at 8 Weeks Post Treatment
Description: Change in baseline subjective fibromyalgia symptoms based on a 100 point scale (0 = no fibromyalgia or minimum score, 100 = severe fibromyalgia and maximal score) from baseline (T=Zero, prior to drug/placebo treatment) to week 8
Time Frame: from baseline to 8 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cyclobenzaprine ER | Placebo
Number analyzed (Participants) | 16 | 12
units on a scale | 59 [36 to 59] | 51 [40 to 51]
Statistical Analysis 1: Comparison: Cyclobenzaprine ER vs Placebo; Test type: Superiority or Other; p = .869, t-test, 2 sided; Mean Difference (Final Values) = 17 — As above- this was the difference between the groups on mean avg, it was used here
Statistical Analysis 2: Comparison: Cyclobenzaprine ER vs Placebo; Test type: Superiority; p = .275, t-test, 1 sided; Mean Difference (Final Values) = 17

ADVERSE EVENTS:
Time Frame: During acute study (8 Weeks)
Groups:
- Placebo: inactive placebo matching
Arm/Group | Cyclobenzaprine ER | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 2/16 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclobenzaprine ER (N=16) | Placebo (N=12)
glucosemia (Endocrine disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
dizziness (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Recruitment was halted as advertisements failed to bring in enough subjects.There were 37 enrollees: some screen failed, never started protocol,lost to follow up, some data not analyzable affording 28 subjects to be included

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No